CLINICAL TRIAL: NCT02883257
Title: Clinical and Biological Markers of Response to Cognitive Behavioural Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Lena Quilty, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003/2016
Record Dates: First submitted 2016-08-19; First posted 2016-08-30 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Depression
Keywords: Major Depression; Major Depressive Disorder; Persistent Depressive Disorder; Cognitive Behavioral Therapy; Biomarkers
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): * 20 individual 60-minute appointments over the course of 16 weeks
  * Consistent with Beck, Rush, Shaw, and Emery (1979)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy will include core mandatory modules of key effective components (e.g., behavioural activation, cognitive restructuring) and optional elements to address individual maintaining factors (e.g., coping and social skills training, perfectionism and self-criticism).

SUMMARY:
The purpose of this study is to locate clinical markers (for example, interviews, questionnaires, and computer tasks) and biological markers (for example, physiological, blood-based, or electroencephalography measurements) that predict response to cognitive behavioral therapy for depression.

DETAILED DESCRIPTION:
Forty adult outpatients with major depressive disorder or persistent depressive disorder will receive up to 20 sessions of cognitive behavioral therapy for depression over 16 weeks. Participants will complete clinical measures (interviews, questionnaires, and computer-based tasks) and biological measures (blood tests, physiological measurements, electroencephalography ) before, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder or Persistent Depressive Disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition
* Must be fluent in English
* Must be capable to give informed consent

Exclusion Criteria:

* Lifetime diagnosis of Schizophrenia, Schizoaffective Disorder, Bipolar Disorder
* Current Alcohol or Drug Use Disorder (except tobacco or caffeine)
* Current psychotic symptoms
* Acute suicide risk
* Psychological treatment for depression initiated during the past three months
* Pharmacological treatment for depression initiated/changed during the past three months
* Previous non-response to two or more adequate trials of pharmacotherapy
* Current significant neurological disorder, head trauma, or unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | 16 weeks
  Depression symptom severity

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (QIDS) | 16 weeks
  Depression symptom severity
World Health Organization Quality of Life Short Version (WHOQOL-BREF) | 16 weeks
  Quality of life
Hamilton Depression Rating Scale (Ham-D) | 16 weeks
  Depression symptom severity
Beck Depression Inventory (BDI) | 16 weeks
  Depression symptom severity
Work and Social Adjustment Scale (WSAS) | 16 weeks
  Functioning and impairment

CONTACTS AND LOCATIONS:
Overall Officials: Lena C Quilty, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones BDM, Levitan RD, Wang W, Uher R, Rotzinger S, Foster JA, Kennedy SH, Farzan F, Quilty LC, Kloiber S. Metabolic variables associated with response to cognitive behavioural therapy for depression in females: A Canadian biomarker integration network for depression (CAN-BIND) study. J Psychiatr Res. 2021 Oct;142:321-327. doi: 10.1016/j.jpsychires.2021.07.031. Epub 2021 Jul 21. PMID 34419752
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca/research
- See also: Information about research by the Canadian Biomarker Integration Network in Depression — http://www.canbind.ca